CLINICAL TRIAL: NCT06549010
Title: A Pilot Study on the Repeatability of a Novel Perimetric Test Administered Via a Virtual Reality Headset.
Brief Title: Perimetric Testing With Virtual Reality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Envision Health Technologies, Inc. (Industry)
Collaborators: Illinois College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: ENV1
Record Dates: First submitted 2024-08-02; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma
Keywords: Glaucoma; Perimetric test; virtual reality
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: 30 healthy subjects 30 glaucoma subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Healthy subjects (Other): 30 healthy subjects
  Interventions: Diagnostic Test: Perimetric test
- Glaucoma subjects (Other): 30 glaucoma patients, 10 mild, 10 moderate, 10 severe
  Interventions: Diagnostic Test: Perimetric test

INTERVENTIONS:
Diagnostic Test: Perimetric test — This study aims to evaluate a novel head-mounted perimeter against the HFA as an alternative method of VF testing. This new perimeter uses a Virtual Reality (VR) headset and a gamified version of VF testing to assess the visual function of healthy eyes and patients.

SUMMARY:
Perimetry is an essential component in the diagnosis and monitoring of glaucoma. Since the advent of Standard Automated Perimetry (SAP), one of the clinical standards has been the Humphrey Field Analyzer (HFA, Carl Zeiss AG, Oberkochen, Germany). Visual field (VF) testing provided by the HFA is standard-of-care in glaucoma clinics and other ophthalmology and optometry practices. However, the HFA is a large device that does not allow for examination outside the clinic and can be uncomfortable for patients with limited mobility.

This study aims to evaluate a novel head-mounted perimeter against the HFA as an alternative method of VF testing. This new perimeter uses a Virtual Reality (VR) headset and a gamified version of VF testing to assess the visual function of healthy eyes and patients. The results of this study will potentially serve as pilot data for the design of a larger study that involves the full assessment of the VR headset and its VF test, based on various testing strategies.

DETAILED DESCRIPTION:
Procedures:

1. Ophthalmic screening:

   (a) Visual acuity, slit lamp exam, rebound tonometry (all subjects)
2. OCT examination of the study eye with the Topcon Maestro2 Optical Coherence Tomography (OCT):

   (a) Standard Retinal Nerve Fiber Layer (RNFL), Optic Disc and Ganglion Cell Complex (GCC) scan patterns (i) Fundus photo is automatically obtained. (b) Abnormalities consistent with ophthalmic disease will be an exclusion for the healthy group of subjects. Reasonable and common artifacts that do not significantly impair the scan report will be accepted.

   (c) OCT abnormalities consistent with glaucoma are expected on the 30 glaucoma subjects.
3. Once eligible, each patient will perform four (4) visual field tests:

   (a) once with the HFA Swedish Interactive Threshold Algorithm (SITA) Standard 24-2 pattern (i) Reliability criteria: False Positives no higher than 15% (b) three tests with the VR headset: (i) two tests with ZEST strategy (ii) one test with gamified ZEST strategy (c) Counter-balancing will be used to determine the order of (a) and (b). In particular, a study participant will either start with the HFA visual field test and then proceed to the three tests with the VR headset; or, start with the three VR tests and finish with the HFA visual field test. The sequence of the visual field tests for each study ID will be provided by the sponsor.

ELIGIBILITY:
Inclusion / Exclusion Criteria:

1. Age range: 25-70 years
2. For normal subjects:

   1. Patient is free of any current or prior ophthalmic pathologies that would potentially cause visual field defects: e.g. retina pathology, glaucoma, cataracts, keratoconus
   2. No ocular surgery other than cataract surgery within 6 months prior to the study visit
3. For glaucoma subjects:

   1. Patient has a diagnosis of primary open-angle glaucoma
   2. Patient is free of any other current or prior ophthalmic pathologies that would potentially cause visual field defects.
   3. No other ocular surgery other than glaucoma or cataract surgery within 6 months prior to the study visit
   4. No IOP lower than 10 mm/Hg or higher than 30 mm/Hg
4. Refractive Error:

   1. Sphere = up to -6.00 D to and up +3.00
   2. Cylinder = up to -3.00 is common
5. No past refractive eye surgery
6. No Multifocal or phakic (ICLs) IOL; no multifocal CLs
7. One eligible eye
8. Ability to sit for standard VF bowl exam. Ability to wear VR perimetry headset device.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Visual field perimetry light sensitivity | 1 day
  Localized differential light sensitivity threshold measured in decibels (dB)
Visual field perimetry foveal sensitivity | 1 day
  Foveal threshold in decibels (dB)
Visual field perimetry test duration | 1 day
  Test duration measured in minutes

SECONDARY OUTCOMES:
Optical Coherence Tomography (OCT) | 1 day
  Optical Coherence Tomography (OCT) thickness values may be used, such as Retinal nerve fiber layer (RNFL) and ganglion cell complex (GCC) thickness, measured in microns.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chaglasian, OD, Principal Investigator — Illinois College of Optometry
Locations (1):
- Illinois College of Optometry / Illinois Eye Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and data analysis will be shared for communication of results and learning conclusions.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will submitted for publication in a medical journal, within 3-6 months of completion of the data analysis of the monitored and locked database.
Access Criteria: The trial results will be published in an open-access medical journal.

REFERENCES:
- [Background] Montesano G, Bryan SR, Crabb DP, Fogagnolo P, Oddone F, McKendrick AM, Turpin A, Lanzetta P, Perdicchi A, Johnson CA, Garway-Heath DF, Brusini P, Rossetti LM. A Comparison between the Compass Fundus Perimeter and the Humphrey Field Analyzer. Ophthalmology. 2019 Feb;126(2):242-251. doi: 10.1016/j.ophtha.2018.08.010. Epub 2018 Aug 14. PMID 30114416
- [Background] Marin-Franch I, Turpin A, Artes PH, Chong LX, McKendrick AM, Alawa KA, Wall M. The Open Perimetry Initiative: A framework for cross-platform development for the new generation of portable perimeters. J Vis. 2022 Apr 6;22(5):1. doi: 10.1167/jov.22.5.1. PMID 35385053
- [Background] Marin-Franch I, Swanson WH. The visualFields package: a tool for analysis and visualization of visual fields. J Vis. 2013 Mar 14;13(4):10. doi: 10.1167/13.4.10. PMID 23492926
- [Background] Bradley C, Ahmed IIK, Samuelson TW, Chaglasian M, Barnebey H, Radcliffe N, Bacharach J. Validation of a Wearable Virtual Reality Perimeter for Glaucoma Staging, The NOVA Trial: Novel Virtual Reality Field Assessment. Transl Vis Sci Technol. 2024 Mar 1;13(3):10. doi: 10.1167/tvst.13.3.10. PMID 38488433